CLINICAL TRIAL: NCT02196428
Title: Medical Telemonitoring Plus Individual Teleconsultation Based on an Ambient Assisted Living (AAL-) Wizard - an Interdisciplinary, Integrated Innovation.
Brief Title: Medical Telemonitoring Plus Individual Teleconsultation in Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: USZ 14809.2
Record Dates: First submitted 2014-07-17; First posted 2014-07-22 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Telemedicine
Keywords: Ambient Assisted Living (AAL); Telemonitoring; Teleconsultation
MeSH Terms: interventions — Remote Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Telemonitoring and Teleconsultation (Other)
  Interventions: Other: Telemonitoring and Teleconsultation

INTERVENTIONS:
Other: Telemonitoring and Teleconsultation — The interventions of this study are supported by a so-called Ambient Assisted Living Wizard (AAL Wizard). This is an IHE-compliant documentation and communication platform with an integrated electronic health record, which enables the study participants (elderly) to manage and store their relevant health data. It includes personal master data and the documentation of telemonitoring data. Additionally, the AAL-Wizard provides the communication modules such as telephone -, video- and time- and online consultation. The tele doctor assess the data (eg, vital signs and content of the medical teleconsultation) and collaborates in this way with the older person, family physicians and other health care providers based on an innovative and flexible telemedical home care service.

SUMMARY:
The aim of this study is to explore the requirements and conditions of medical teleconsultation and remote diagnostics (telemonitoring) of older people in the residential environment with an emphasis on the need for adaptation, feasibility and acceptance of telemedicine services to a web based documentation and communication platform (Ambient Assisted Living Wizard).

DETAILED DESCRIPTION:
The technical development of the so-called "AAL Wizard" is basis for the study. The AAL-Wizard is an IHE(Integrating the Healthcare Enterprise)-compliant, web based documentation and communication platform with an integrated electronic patient record, which can be used by the study participants during the study. Vital parameters are collected with the help of certified medical products according to the guidelines "93/42/EEC(European Economic Community) on medical devices" (e.g. blood pressure devices, scales, pedometers), transmitted electronically, documented and archived directly in the system. Vital parameters out of range will be prioritized displayed in the AAL Wizard (e.g. traffic light system, short message notification, pop-up function, etc.) and the study participant will be contacted by the tele doctor (teleconsultation) . The decision on the necessary intervention (e.g. contact of the in-house home care, therapeutic and diagnostic recommendations or recommendation of a primary care consultation /hospital submission) are in the responsibility of the tele doctor based on the communication with the patient and the family doctor's recommendations for the treatment of his patient.

At the beginning of the study, the tele doctors of the Clinical Telemedicine at the University Hospital Zurich (USZ) perform an appointment with the respective study participants. The electronic patient record will be set up and the process of the telemonitoring will be defined.

ELIGIBILITY:
Inclusion Criteria:

* german speaking
* voluntary participation
* written consent of the trial participant after enlightenment

Exclusion criteria:

* apply to health conditions (physical and / or psychological) when verbal communication and / or the operation of the AAL Wizard and an independent living in their own living area is not possible.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
User profile of medical telemonitoring and teleconsultation | 10 months
  Objective criteria:
  Age, sex, weight, height, education, civil status, diagnosis, medical history, medication, alcohol and tabacco consumption using interval, nominal and ordinal scales.
  Subjective criteria:
  1. Subjective state of health : German questionnaire Short Form (SF)-36/SF-12
  2. Integration into social networks and assessment of social support, self-management skills: 10-item questionnaire using 5-point Likert scale responses do not apply at all (1) to apply (5).
  3. Health literacy: 13-item questionnaire using 4-point Likert scale responses do not apply (1) to apply (4).
Demand of health information | 10 months
  Text analysis with inductive category developement of teleconsultation services via telephone, video and online consultation and telemonitoring
Acceptance medical telemonitoring and teleconsultation | 10 months
  1. Observed acceptance in relation to the intervention
     * compliance using inducive category development
     * quality of service : 3-item questionnaire using 5-point Likert scale responses do not apply at all (1) to apply (5)
  2. Acceptance of user using inducive category development

SECONDARY OUTCOMES:
Acceptance and demand of health information of secondary end users of telemedical services | 10 months
  Acceptance and demand of health information of telemedical service of secondary end users (family practitioner, other caregivers, family) using text analysis with inductive category developement and open structured, inductive questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Brockes, MD, PD, Principal Investigator — University Hospital Zurich, Rämistrasse 100, 8091 Zurich, Switzerland
Locations (1):
- Clinical Telemedicine, University Hospital Zurich, Zurich, Canton of Zurich, Switzerland